CLINICAL TRIAL: NCT05521945
Title: Effect of Intermittent Fasting on Body Composition, Clinical Health Markers and Memory Status Among Adult Population: A Randomized Control Trial
Brief Title: Effect of Intermittent Fasting Among Adult Population
Acronym: IF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Punjab (Other)
Responsible Party: Principal Investigator, Zahara Ali Rizvi, principal investigator, University of the Punjab
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZAHARA ALI RIZVI
Record Dates: First submitted 2022-08-10; First posted 2022-08-30 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Intermittent Fasting
Keywords: Intermittent fasting; Memory status; physical activity; customized diet plan; 24- hour dietary recall; Multifactorial Memory Questionnaire
MeSH Terms: conditions — Intermittent Fasting; Motor Activity | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intermittent Fasting Group (Experimental): eight hours eating window and 16 hours for fasting among healthy population
  Interventions: Behavioral: Intermittent Fasting
- Customized Dietary group (Active Comparator): Customized diet plan according to participants' calorie intake and according to their respective Body Mass Index
  Interventions: Behavioral: Calorie Restricted Diet
- Control group (Placebo Comparator): Normal routine diet
  Interventions: Behavioral: Normal dietary intake

INTERVENTIONS:
Behavioral: Intermittent Fasting — 16 hours fasting and 8 hours eating window
  Arms: Intermittent Fasting Group
Behavioral: Calorie Restricted Diet — The customized diet plan will be given to the participants according to their calorie intake requirements
  Arms: Customized Dietary group
Behavioral: Normal dietary intake — normal diet without any customization
  Arms: Control group

SUMMARY:
Our study aims to assess the effects of intermittent fasting among the healthy population.

DETAILED DESCRIPTION:
Research needs to be conducted to find the effects of intermittent fasting on humans as it might not have the same favorable effects on the memory of a human brain compared to mice. This study will also help to assess the consequences of different intermittent fasting regimens on different individuals (based on age, sex, body mass index , memory status and physical activity etc)

ELIGIBILITY:
Inclusion Criteria:

* BMI greater or equal to 25kg/m2.

Exclusion Criteria:

not given consent having secondary or syndromic forms of obesity taking medication for weight gain or reduction undergoing bariatric surgery

* diabetic pregnant women breastfeeding mothers chronic disease

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Weight(in kg) | three months
  For BMI
Height (in cm) | three months
  for BMI
Waist (in cm) | three months
  for waist hip ratio
Hip measurement(in cm) | three months
  for waist hip ratio

SECONDARY OUTCOMES:
Clinical Health Markers | three months
  Low Density Lipid, Very Low Density Lipid, High Density Lipid, triglycerides
blood sugar | three months
  Fasting blood sugar level
blood pressure | three months
  Diastolic and systolic blood pressure

OTHER OUTCOMES:
Memory Status | three months
  scoring system higher the value good will be results

CONTACTS AND LOCATIONS:
Overall Officials: Javeria Saleem, Ph.D, Study Director — University of the Punjab
Locations (1):
- University of the Punjab, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
participants assessment report regarding intermittent fasting

REFERENCES:
- [Derived] Rizvi ZA, Saleem J, Zeb I, Shahzad R, Kayani JA, Faryal J, Bukhari GMJ, Abdi G, Jain M. Effects of intermittent fasting on body composition, clinical health markers and memory status in the adult population: a single-blind randomised controlled trial. Nutr J. 2024 Nov 28;23(1):147. doi: 10.1186/s12937-024-01046-9. PMID 39609683